CLINICAL TRIAL: NCT07004179
Title: Implementation of a Diabetic Foot Prevention Strategy in Primary Care: Study Protocol for Two-arm Cluster Randomised Controlled Trial (iMplanta Study)
Brief Title: Implementation of a Diabetic Foot Prevention Strategy in Primary Care (iMplanta Study)
Acronym: iMplanta
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Collaborators: Universitat de les Illes Balears (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PI06_2024
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Disease; Diabetic Foot Ulcer (DFU)
Keywords: Diabetic foot; Implementation Sciencie; Prevention; Primary Care
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implementation Mapping strategy (Experimental): Primary care centers, participants and caregivers assigned to this group will be part of an intervention designed to adopt an implementation strategy that will enhance the effective integration of the Diabetic Foot Care Protocol by reducing the complications associated with diabetic foot.
- Current implementation strategy for diabetic foot prevention (Sham Comparator): Primary care centers, along with the participants and caregivers assigned to this group, will be integrated into routine care to prevent complications associated with diabetic foot.
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Behavioral: Implementation strategy developed using the Implementation Mapping model to enhance the effective integration of the Protocol for Assistance to People with Diabetic Foot — The intervention will be based on the Implementation Mapping methodology (IM). This model is based on the Intervention Mapping. IM consists of several specific tasks:
  1. Conduct an assessment of needs and identification of programme adopters and implementers through a review of qualitative or mixed studies assessing the perceptions of both patients and professionals regarding DF prevention as well as individual semi-structured interviews with patients, health professionals and management staff
  2. Indicate adoption and implementation outcomes and action objectives, identifying determinants and create matrices of change; this process will allow for the identification of determinants, which are those factors that influence the actions will be implemented
  3. Select theoretical methods and select or design implementation strategies using the ERIC model (Expert Recommendations for Implementing Change)
  4. Produce implementation protocols and materials
  5. Evaluate implementation results
Other: Sham Comparator — Usual care: No systematic implementation of the protocol based on the prevention of foot at risk, ulcer treatment and screening of the risk of diabetic foot ulcer for referral to hospital care.
  Arms: Current implementation strategy for diabetic foot prevention

SUMMARY:
The goal of this two-arm cluster randomised controlled trial (RCT) is to evaluate the effectiveness of a new implementation strategy based on the ImM model for the Protocol of assistance to the person with diabetic foot (PAPDF) of the Balearic Islands Health Service in reducing complications of diabetic foot, compared to the current implementation strategy, in the primary care centers of Majorca. As secondary objectives we aim 1. To determine the reach of the implementation strategy in the GAPM primary care centers, 2.To compare the effectiveness of the PAPDF versus usual care in preventing diabetic foot complications, 3. To identify the number of healthcare professionals adhering to the implementation strategy and 4. To assess the sustainability of the implementation strategy over time.

DETAILED DESCRIPTION:
A two-arm, cluster-randomized clinical trial will be conducted. The unit of randomization will be the primary care centers (PCCs) within the Mallorca Primary Care Management (GAPM). The PCCs will be randomly assigned to the intervention group, that will apply an implementation strategy based on the Implementation Mapping (ImM) model and the control group, that will receive no specific intervention, and the implementation of the PAPDF will continue as currently practiced in the participating PCCs.

Data collection will be carried out at baseline (visit 0), at six months (visit 1), and 12 months (visit 2) for follow-up.

Four primary care centers (PCCs) will be included in the study. Since the implementation of the PAPDF intervention will be integrated into the routine care of the participating PCCs, all healthcare professionals working in the selected centers will be automatically included in the study. Patients from the PCCs meeting the following criteria will be eligible for participation: Diagnosis of type 1 or type 2 diabetes mellitus (DM), aged 18 years or older, attending nursing consultations at participating PCCs during the study period. To assess the occurrence of complications associated with PD, cross-sectional samples of patients with DM in the selected health centres will be selected at different time points: before implementation (baseline), which will correspond to data from the 12 months prior to the start of the study, and at 6 and 12 months after the start of the study.

Eligible participants will be patients with a diagnosis of type 1 and 2 DM, over 18 years of age, who belong to the Public Health Service of the Balearic Islands of one of the selected centres. Will be excluded individuals with gestational diabetes, patients with DF ulcers or lower limb amputations prior to the start of the study.

The selected health centres will be randomly distributed into the control or intervention group using a computerised randomisation tool. Due to the characteristics of the implementation intervention, blinding will not be possible. However, there will be blinding for the team responsible for data analysis, as they will not know to which randomisation group (control/intervention) the data will belong.

The intervention will be based on the Implementation Mapping methodology. This model is based on the Intervention Mapping, which is step 5 of the model. In turn, ImM consists of several specific tasks: 1) conduct a needs assessment and identification of programme adopters and implementers; 2) indicate adoption and implementation outcomes and action objectives, identify determinants and create matrices of change; 3) select theoretical methods and select or design implementation strategies; 4) produce implementation protocols and materials; 5) evaluate implementation results.

1. In order to carry out the implementation needs assessment, this task will be developed in two phases:

   1.1. Review of available evidence. A review of qualitative or mixed studies assessing the perceptions of both patients and professionals regarding the prevention of DF has been carried out in order to identify possible barriers and facilitators that could be useful for implementation in our context.

   1.2. Identification of implementation needs in the context of the project: In order to find out the specific needs of the agents involved at the different levels of our context, data collection and analysis will be carried out using qualitative research methods. First of all, individual semi-structured interviews will be conducted with DM patients, health professionals (nurses, doctors, podiatrists) and management staff of the GAPM. In order to approach the context under study, the categories have been established taking into account the geographical distribution of the 47 health centres on the island of Mallorca, according to the health sector to which they belong: Ponent, Migjorn, Llevant or Tramuntana sectors. In addition, the different geographical areas have been taken into account, as the needs may be different depending on whether the health sector is rural or urban.

   Regarding the health professionals involved, priority will be given to recruiting nurses, as they are the ones who carry out DF screening in PCC in our area and doctors who work with a quota of adults in a GAPM health centre, and who are active at the time the study is carried out. 4 podiatrists who currently exist on the island of Mallorca belonging to the Health Service of the Balearic Islands, as they are considered a key figure in the development of DF care. Management personnel will also be selected to carry out organizational tasks in the GAPM during the development of the project.

   In addition, focus groups will be conducted with participants from the 3 categories (patients, professionals and staff of the organisation).

   Initially, 20 participants will be recruited for interviews and focus groups selected through purposive sampling, although this number may increase or decrease depending on when the theoretical saturation of the data collected is reached.

   The recruitment of healthcare professionals will be carried out via corporate mail Office 365 Ib-Salut, which will briefly explain the objectives of the study and the necessary involvement of the participants. An email address and a contact telephone number will be provided so that potential participants can obtain additional information or clarify any doubts. If they finally decide to participate in this phase of the study, participants should contact the research team, who will provide them with the information sheet and informed consent.

   As for patients, recruitment will be done through the health professionals of the health centre, who will offer the possibility of participating in the project and will provide basic information and contact details of the research team. Information posters about the project will also be placed in the participating health centres. They will also be given the information sheet and the informed consent form. In case the minimum required sample is not reached, snowball recruitment will be carried out.

   To facilitate qualitative data collection, these interviews will be conducted according to the Consolidated Framework for Implementation Research (CFIR) construct-based interview guide. Interviews and focus groups will be recorded via audio recorder and then transcribed for analysis. Data analysis (content analysis) will also be carried out using the CFIR framework to facilitate further interpretation of the data and its direct application in the implementation process. In addition, the qualitative data analysis software Atlas.ti will be used.
2. Identification of adoption and implementation outcomes, action targets, determinants and change targets.

   These outcomes refer to those objectives that the implementation intervention is intended to achieve. This process will allow for the identification of determinants, which are those factors that influence whether or not the actions will be implemented.

   The IM model proposes to develop matrices that combine action objectives and determinants to propose change objectives. These matrices will need to be adapted to the specific needs of the implementation context as identified through interviews and focus groups.

   The change objectives are the necessary transformations to be carried out in order to achieve the proposed results.
3. Select theoretical methods and select or design implementation strategies:

   This phase aims to act on the determinants previously identified based on theoretical methods designed for this purpose. In addition, the design of context-specific implementation strategies will be carried out.

   As a theoretical framework, the ERIC model (Expert Recommendations for Implementing Change) has been selected. This is a compilation of 73 implementation strategies that allows for the selection of interventions to guide the implementation process.

   A combination of ERIC- CFIR models will be used to facilitate the selection of implementation strategies based on the results of the context analysis conducted in Task 2.

   In addition, behavioural change models will be used to influence changes at the individual level increasing knowledge, improving risk perception, modifying attitudes and beliefs, increasing self-efficacy, improving skills, etc. The use of Social Cognitive Theory is proposed to address personal determinants.
4. Produce implementation protocols and materials:

   The production of specific implementation materials, derived from all the work done in the previous tasks, will be carried out. For this task, representatives of all the parties involved (patients with DM, health professionals (physicians, nurses, podiatrists) and GAPM management staff) will be involved in the creation of the final material.
5. Evaluate implementation results:

This task will be developed using the RE-AIM model which is based on the evaluation of 5 outcome dimensions: reach, effectiveness, adoption, implementation and maintenance. The interactive online tool available on the RE-AIM website ( https://re-aim.org ) will be used. An indicator will be assigned to each dimension:

Reach- Percentage of DM patients meeting inclusion criteria exposed to the PAPDF in both groups.

Effectiveness- Prevalence of PD ulcers among patients over 18 years of age with DM in both groups.

Adoption- Percentage of nurses who have completed the PD protocol in both groups.

Implementation- Degree of fidelity of implementation of the PAPDF in both groups.

Maintenance- Measured through the Provider REport of Sustainment Scale (PRESS) in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 or type 2 diabetes mellitus.
* Aged 18 years or older.
* Attending nursing consultations at participating primary care centers during the study period.

Exclusion Criteria:

* Patients with gestational diabetes.
* Patients with diabetic foot ulcers prior to the start of the study.
* Patients with lower limb amputations prior to the start of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1520 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Reach | At baseline, 6 months and 12 months.
  Percentage of patients with diabetes mellitus over 18 years of age who have the "Diabetic Foot Protocol" open in the electronic medical record divided by the total number of patients with DM over 18 years of age in the health centers of both groups.

SECONDARY OUTCOMES:
Effectiveness | At baseline, 6 months and 12 months.
  Comparison of the prevalence of diabetic foot ulcers among patients older than 18 years with diabetes mellitus in both groups.
  As a secondary outcome, the prevalence of total lower limb amputations in DM patients older than 18 years will also be compared between the intervention group and the control group.
Adoption | At baseline, 6 months and 12 months.
  Percentage of nurses who have performed the Diabetic Foot Protocol out of the total number of nurses in the center in both groups.
Implementation fidelity | At baseline, 6 months and 12 months.
  Degree to which the implementation of the Diabetic Foot Protocol is delivered as intended in both groups.
  The number of completed protocols will be determined with respect to the total number of open protocols. A completed protocol will be understood as one in which all items have been recorded.
Maintenance | At baseline, 6 months and 12 months.
  Measured through the Provider REport of Sustainment Scale (PRESS) in both groups. This validated scale consists of 3 items that are assessed on a Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Gerència d'Atenció Primària de Mallorca, Palma De Mallorca, Balearic Islands 07002, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No